CLINICAL TRIAL: NCT05564182
Title: Efficacy of High Intensity Laser Treatment in Hemiplegic Shoulder Patients
Brief Title: High Intensity Laser Therapy in the Treatment of Hemiplegic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nur Doğanlar, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HILT2022
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Pain; Hemiplegia; Arthralgia; Joint Diseases; Musculoskeletal Diseases
Keywords: hemiplehic shoulder pain; rotator cuff tear; high intensity laser therapy; exercise; ultrasound
MeSH Terms: conditions — Shoulder Pain; Hemiplegia; Arthralgia; Joint Diseases; Musculoskeletal Diseases; Rotator Cuff Injuries; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity laser therapy + exercise (Experimental): HILT will be applied to the patients five times a week for a period of three weeks and one session per day for a total of 15 sessions by a physical therapy technician who is experienced in using a laser device. (BTL-6000 high intensity laser 12 W, Stevenage, Hertfordshire, England). The laser device generates a maximum power of 12 W and emits a wavelength of 1064 nm (Nd: YAG laser). In the HILT group, it will be used in the rotator cuff muscles area in two stages, Phase I and Phase II. For analgesic effect in phase I. Phase II will also be applied for the biostimulation effect. Exercise program was applied in five sessions a week for three weeks, with a total of 15 sessions a day.
  Interventions: Device: High intensity laser therapy; Other: Therapeutic Exercise
- Exercise only (Active Comparator): Exercise program was applied in five sessions a week for three weeks, with a total of 15 sessions a day.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Device: High intensity laser therapy — HILT will be applied to the patients five times a week for a period of three weeks and one session per day for a total of 15 sessions by a physical therapy technician who is experienced in using a laser device (BTL-6000 high intensity laser 12 W, Stevenage, Hertfordshire, England). It will be used in the rotator cuff muscles area in two stages, Phase I and Phase II. For analgesic effect in phase I. Phase II will also be applied for the biostimulation effect.
  Arms: High intensity laser therapy + exercise
Other: Therapeutic Exercise — Therapeutic Exercise As therapeutic exercise program; A multidisciplinary stroke rehabilitation program will be implemented in the presence of a specialist physiotherapist. In addition, a therapeutic exercise program including passive, actively supported and active ROM exercises, stretching, strengthening and mobilization exercises will be applied to all patients by physiotherapists according to the level of pain and limitation.It was planned to implement a total of 15 sessions 5 days a week for 3 weeks, for approximately 30 minutes.

SUMMARY:
High intensity laser therapy (HILT) has been considered as a treatment option for shoulder pain. In randomized controlled studies with high-intensity laser therapy (HILT), there are publications showing its effectiveness in conditions such as shoulder pathologies such as subacromial impigment syndrome and adhesive capsulitis. However, there are few studies in the literature that focus on the effectiveness of HILT, especially in hemiplegic shoulder pain. In this study, we intended to investigate the effectiveness of HILT on pain, disability, function and quality of life in patients with HSP accompanied by PTRCT.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. Patients with HSP accompanied by PTRCT (n=40) were randomly assigned to HILT and control groups. Group 1 (HILT group, n=20) received 3 sessions of HILT per week for 3 weeks in addition to the exercise program which performed 5 sessions per week for 3 weeks. Group 2 (Control group, n=20) received an exercise program for HSP of 5 sessions per week for 3 weeks.

Participants were evaluated with Visual Analog Scale (VAS), passive Range of Motion (ROM), Shoulder Pain and Disability Index (SPADI), Nottingham Health Profile (NHP), Functional Independence Measure (FIM) and ultrasonographic PTRCT size,Fugl Meyer Assessment, Brunnstrom Stages, Modified Ashworth Scale (MAS) Nottingham Health Profile (NHP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with HSP aged 50-85 years with hemiplegia duration> 2 months, suffered a stroke resulting in unilateral hemiplegia for the first time

Exclusion Criteria:

* Cases who had inflammatory rheumatic disease, cervical radiculopathy, diabetes mellitus, thyroid disease, coronary heart disease, cardiac pace-maker, neurological disease, shoulder surgery, and shoulder injection in the last 3 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Through study completion, an average of 3 weeks (Change from baseline hemiplegic shoulder pain of the patients at 3 weeks
  Severity of pain was assessed using the standart 10 cm VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end

SECONDARY OUTCOMES:
Range of motion (ROM) of the hemiplegic shoulder | Time Frame: Through study completion, an average of 3 weeks (Change from baseline hemiplegic shoulder ROM of the patients at 3 weeks
  Passive ROM measurements of shoulder external rotation, abduction, and flexion movements were recorded by a universal goniometer.
Shoulder Pain and Disability Index (SPADI) | Through study completion, an average of 3 weeks (Change from baseline hemiplegic arm motor recovery of the patients at 3 weeks
  The SPADI is a joint-specific measure focusing on pain and functional activities involving the shoulder.SPADI is self-administered questionnaire composed of 5 items assessing pain and 8 items assessing disability. The score varied from 0% to 100%, with higher scores reflected greater pain and disability
Spastisity | Through study completion, an average of 3 weeks (Change from baseline hemiplegic arm spasticity of the patients at 3 weeks
  The five-point Modified Ashworth Scale (MAS), a clinical scale ranging from 0 to 4 (0 being normal muscle tone, and 4 being rigid) was used for measuring spasticity and muscle tone. Higher scores indicate severe spasticity.
Functional status (FIM) | Through study completion, an average of 3 weeks (Change from baseline functional status of the patients at 3 weeks
  FIM is a universal assessment tool consisting of a total of 18 items that explores an individual's several physical and social functions, such as self-care, transfer, locomotion, sphincter control, communication and social cognition. Each item is scored on a 7-point ordinal scale ranging from complete independence (score= 7) to complete dependence (score= 1). Higher FIM scores indicate higher levels of independence
Quality of life of the hemiplegic patient | Through study completion, an average of 3 weeks (Change from baseline quality of life of the patients at 3 weeks
  Nottingham Health Profile (NHP), a life quality test, includes 38 yes / no statements regarding pain, physical mobility, emotional reactions, sleep, social isolation and energy level. Ratings on each component are weighted to give a score between 0 and 100. Higher NHP scores show a higher level of trouble
Fugl Meyer Assessment (upper extremity) | Through study completion, an average of 3 weeks (Change from baseline quality of life of the patients at 3 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.The FM scale is divided into 5 areas: motor function, sensory function, balance, range of motion, and joint pain. Each domain contains multiple items, each scored on a 3-point ranking scale (0 = unable to perform, 1 = partially performs, 2 = fully performs).Higher scores is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viana R, Pereira S, Mehta S, Miller T, Teasell R. Evidence for therapeutic interventions for hemiplegic shoulder pain during the chronic stage of stroke: a review. Top Stroke Rehabil. 2012 Nov-Dec;19(6):514-22. doi: 10.1310/tsr1906-514. PMID 23192716
- [Background] Tao W, Fu Y, Hai-Xin S, Yan D, Jian-Hua L. The application of sonography in shoulder pain evaluation and injection treatment after stroke: a systematic review. J Phys Ther Sci. 2015 Sep;27(9):3007-10. doi: 10.1589/jpts.27.3007. Epub 2015 Sep 30. PMID 26504346
- [Background] Song HJ, Seo HJ, Lee Y, Kim SK. Effectiveness of high-intensity laser therapy in the treatment of musculoskeletal disorders: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Dec;97(51):e13126. doi: 10.1097/MD.0000000000013126. PMID 30572425